CLINICAL TRIAL: NCT06676735
Title: Research on Intraoperative Hypothermia Risk Prediction and Temperature Management Strategies in Elderly Patients: Construction of Intraoperative Hypothermia Prediction Model Based on Dynamic Incremental Training and Evaluation of Clinical Application Effectiveness
Brief Title: Research on Intraoperative Hypothermia Risk Prediction Model and Temperature Management Strategy for Elderly Patients During Surgery Based on Dynamic Incremental Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Min Su, Director, First Affiliated Hospital of Chongqing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZZ2024-173-01
Record Dates: First submitted 2024-10-31; First posted 2024-11-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Intraoperative Hypothermia
Keywords: Intraoperative hypothermia; Prediction model; Elderly patients; Active warming; Machine Learning

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intraoperative hypothermia low risk group (Experimental): Patients included this group are determined by prediction model. Operating room environment temperature was set at not less than 21°C, with a relative humidity of 50% to 60%. Patients are covered from neck to feet with a cotton blanket and the area to be disinfected and operated on is uncovered after induction of anesthesia. All patients will be administered intravenous fluid warmers and irrigation fluid prewarming (37℃~43℃).
  Interventions: Diagnostic Test: Prediction of intraoperative hypothermia risk; Other: Measurement of tympanic membrane temperature
- Intraoperative hypothermia high risk group (Experimental): Patients included this group are determined by prediction model. In addition to the measures taken in intraoperative hypothermia low risk group, an inflatable warming system, including a forced air warming system and forced air warming blanket, is employed for prewarming before anesthesia initiation and for maintaining body temperature throughout the operation. During the surgery, the insulation blanket will be applied to non surgical areas, and the host temperature will be adjusted to 38 ℃ for warming. If the temperature of the patient is lower than 36 ℃, the temperature of the system can be adjusted to 43 ℃; if the temperature of the patient is higher than 37 ℃, the temperature of the system can be adjusted to 32 ℃. After the patient's temperature is normal, it can be adjusted back to 38 ℃.
  Interventions: Device: Inflatable warming system; Diagnostic Test: Prediction of intraoperative hypothermia risk; Other: Measurement of tympanic membrane temperature
- Model optimization group (Other): Only observe the patient's baseline, intraoperative hypothermia, postoperative complications, and other indicators, and collect data through the electronic Data Capture System to optimize existing intraoperative hypothermia prediction model. The estimated sample size is 600 cases by the incremental learning curve calculating.
  Interventions: Other: The difference between axillary temperatature and core temperature in elderly patients; Other: Measurement of tympanic membrane temperature
- Group of model benefit evaluation (No Intervention): Data of this group is medical records before the application of the intraoperative hypothermia prediction model, which will be collected from the electronic medical record system.

INTERVENTIONS:
Device: Inflatable warming system — Inflatable warming system, including a forced air warming system (IOB, WU505) and forced air warming blanket (IOB-001, IOB-006, IOB-011), is employed for prewarming before anesthesia initiation and for maintaining body temperature throughout the operation. During the surgery, the insulation blanket will be applied to non surgical areas, and the host temperature will be adjusted to 38 ℃ for warming. If the temperature of the patient is lower than 36 ℃, the temperature of the system can be adjusted to 43 ℃; if the temperature of the patient is higher than 37 ℃, the temperature of the system can be adjusted to 32 ℃. After the patient's temperature is normal, it can be adjusted back to 38 ℃.
  Arms: Intraoperative hypothermia high risk group
Diagnostic Test: Prediction of intraoperative hypothermia risk — According to the Intelligent Care For The Elderly (ICE, an optimized model based on the existing prediction model of our research group after dynamic incremental training), patients are divided into intraoperative hypothermia lowrisk group and intraoperative hypothermia high risk group.
  Arms: Intraoperative hypothermia high risk group; Intraoperative hypothermia low risk group
Other: The difference between axillary temperatature and core temperature in elderly patients — Previous studies have shown that the difference and standard deviation between esophageal temperature and axillary temperature are core 0.05 ℃ and 0.26 ℃, respectively. In light of 10% dropout rate, a integer sample size of 400 achieves 95% power to detect a mean of paired differences of 0.05 with an estimated standard deviation of paired differences of 0.26 and with a significance level (alpha) of 0.05 using a two-sided paired t-test. So 400 patients in the Model optimization group need to undergo core temperature (esophageal temperature or nasopharyngeal temperature).
  Arms: Model optimization group
Other: Measurement of tympanic membrane temperature — As a intraoperative core temperature reference (measure every 15 minutes) for patients without esophageal temperature or nasopharyngeal temperature monitoring.
  Arms: Intraoperative hypothermia high risk group; Intraoperative hypothermia low risk group; Model optimization group

SUMMARY:
With the support of partial dual temperature monitoring (comparing the specific difference between standardized axillary temperature monitoring and esophageal temperature), this trial is divided into the following three parts:

1. Multi center observational study: Establish and validate a dynamic incremental training intraoperative hypothermia prediction model - Intelligent Care for the Elderly (ICE) - Intraoperative hypothermia warning system, and provide ICE Offline for use by healthcare professionals and ICE Online for further model updates when needed for clinical or research purposes.
2. Multi center non randomized controlled clinical trial: Conduct a multi center stratified temperature management clinical trial based on ICE Offline after dynamic incremental training to verify the clinical and economic benefits of the model and active warming.
3. Pre and post comparative study: Collect data before ICE application and compare it with data after ICE promotion.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (aged 60 and above) undergoing non cardiac elective surgery under general anesthesia;
* 30 minutes ≤ Estimated surgical duration ≤ 240 minutes ;
* Normal preoperative bleeding and clotting time
* American society of Aneshesiologists physical status classification system:Ⅰ～Ⅳ

Exclusion Criteria:

* Mental illness
* Cirrhosis
* Existence or potential central hyperthermia
* Metabolic thermoregulatory abnormalities
* History of malignant hyperthermia or family history
* Extensive skin burns or injuries
* Seriously infect
* Long term use of nonsteroidal anti-inflammatory drugs
* Expected difficult airway
* Researchers believe that individuals who are not suitable to participate in clinical trial
* Refusal to sign informed consent form
* Withdraw informed consent form
* Severe bleeding or shock during perioperative period.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1323 (Actual)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-01-14 (Actual)

PRIMARY OUTCOMES:
Intraoperative hypothermia | Up to 24 hours, from the time of entry into the operating room to the time of exit from the operating room.
  Intraoperative hypothermia, defined as a core temperature below 36 °C

SECONDARY OUTCOMES:
The specificity and sensitivity of the model | 1 year
  Conventional parameters for evaluating model accuracy
Physical sensation | Perioperative period
  The ASHRAE thermal sensation scale, which was developed for use in quantifying people's thermal sensation, is defined as follows:+3 (hot), +2 (warm), +1 (slightly warm), 0 (neutral), -1 (slightly cool), -2(cool), and -3 (cold)
Total volume of intraoperative blood loss | Intraoperative
  Routine intraoperative monitoring indicators
Postoperative shivering | Up to 60 minutes
  A compensatory response of the body to hypothermic stimuli that cause rapid rhythmic. Once the operation is completed, the patient will be extubated and the presence or absence of shivering will be recorded up to 60 minutes after the extubation with the Badjatia 2008 scale consisting of a gradual evaluation of 0 to 3 points. With scores greater or equal to 1, shivering is considered established.
Postoperative coagulation index | Within 24 hours after operation
  Routine postoperative monitoring indicators
Postoperative hospital stay | Through study completion, an average of 1 year
  The number of days from the end of surgery to discharge displayed in the electronic medical record system for patients
Total hospital stay | Through study completion, an average of 1 year
  The number of days from admission to discharge displayed in the electronic medical record system for patients.
Costs of using active warming | Perioperative period
Postoperative hospital costs | Through study completion, an average of 1 year
  The Postoperative hospital cost (￥) from the end of surgery to discharge displayed in the electronic medical record system
Total hospital costs | Through study completion, an average of 1 year
  The Total hospital cost (￥) from admission to discharge displayed in the electronic medical record system
30-day postoperative readmission | 30 days after operation
  Routine postoperative monitoring indicators
30-day postoperative complications | 30 days after operation
  Routine postoperative monitoring indicators
30-day postoperative mortality | 30 days after operation
  Routine postoperative monitoring indicators
Heart rate | Perioperative period
  Obtained from multi parameter monitor
Blood pressure | Perioperative period
  Obtained from multi parameter monitor
Blood oxygen saturation | Perioperative period
  Obtained from multi parameter monitor

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data Data available: Yes Data types: Identified participant data How to access data: atpcr7@yeah.net When available: Within 5years after this trial
  Supporting Documents Document types: None
  Additional Information Who can access the data: Researchers whose proposed use of the data have been approved by Leader Sponsor and Principal Investigator of this trial.
  Types of analyses: To be discussed with the steering committee. Mechanisms of data availability: With investigator support after approval signed data access agreement.
  Any additional restrictions: None
Supporting Information: Study Protocol, SAP, CSR